CLINICAL TRIAL: NCT00017147
Title: A Phase III Study of Radiation Therapy (RT) and O6-Benzylguanine (O6-BG) Plus BCNU Versus RT and BCNU Alone for Newly Diagnosed Glioblastoma Multiforme (GBM) and Gliosarcoma
Brief Title: S0001 RT and Carmustine With or Without O6BG in Patients With New Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068656; S0001 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Malignant Neoplasms of Eye, Brain and Other Parts of Central Nervous System
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Carmustine; Radiotherapy; O(6)-benzylguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- O6-BG + BCNU + Radiation Therapy (Experimental): O6-BG: 120 mg/m^2 IV over 1 hour on day 1 of each cycle BCNU: 40 mg/m^2 IV over 1 hour on day 1 of each cycle 6 hours after O6-BG dose. Radiation Therapy: 5 days/week using one fraction per day and a dose of 180 cGy per fraction. Initial target volume is dose of 5040 cGy in 28 fractions with boost target volume of 1080 cGy in 6 fractions.
  Interventions: Drug: carmustine; Radiation: radiation therapy; Drug: O6-Benzylguanine
- BCNU + Radiation Therapy (Active Comparator): BCNU: 40 mg/m^2 IV over 1 hour on day 1 of each cycle. Radiation Therapy: 5 days/week using one fraction per day and a dose of 180 cGy per fraction. Initial target volume is dose of 5040 cGy in 28 fractions with boost target volume of 1080 cGy in 6 fractions.
  Interventions: Drug: carmustine; Radiation: radiation therapy

INTERVENTIONS:
Drug: carmustine — 40 mg/m^2 IV over 1 hour on day 1 of each cycle 6 hours after O6-BG dose for experimental arm with O6=BG.
  200 mg/m^2 IV over 1 hour on day 2 of each cycle for the active comparator arm.
Radiation: radiation therapy — 5 days/week using one fraction per day and a dose of 180 cGy per fraction. Initial target volume is dose of 5040 cGy in 28 fractions with boost target volume of 1080 cGy in 6 fractions.
Drug: O6-Benzylguanine — 120 mg/m^2 IV over 1 hour on day 1 of each cycle
  Other Names: O6-BG
  Arms: O6-BG + BCNU + Radiation Therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. O6-benzylguanine may help carmustine kill more tumor cells by making tumor cells more sensitive to the drug. It is not yet known whether radiation therapy and carmustine are more effective with or without O6-benzylguanine.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus carmustine with or without O6-benzylguanine in treating patients who have newly diagnosed glioblastoma multiforme or gliosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival, failure-free survival, and progression-free survival of patients with newly diagnosed glioblastoma multiforme or gliosarcoma treated with radiotherapy and carmustine with or without O6-benzylguanine.
* Compare the frequency and severity of toxic effects of these regimens in these patients.
* Correlate the survival of these patients with the expression of O6-alkylguanine-DNA alkyltransferase.

OUTLINE: This is a randomized study. Patients are stratified according to age (under 50 vs 50 and over), prior surgery (biopsy only vs resection), and Zubrod performance status (0-1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy daily 5 days a week over 7 weeks for a total of 34 fractions. Patients also receive chemotherapy comprising O6-benzylguanine IV over 1 hour followed 6 hours later by carmustine IV over 1 hour on day 1 of radiotherapy. Chemotherapy repeats every 6 weeks for a maximum of 7 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo radiotherapy as in arm I. Patients receive carmustine IV as in arm I.

Patients are followed at week 48, every 4 months for 1 year, and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 375 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme or gliosarcoma

  * Biopsy or surgical resection within the past 28 days

    * MRI* with gadolinium performed before registration
    * Patients who undergo a simple biopsy only require preoperative MRI* with gadolinium
* No more than 2 noncontiguous tumor sites based on T2-weighted MRI (in 3 dimensions)*
* No prior radiotherapy-delivered cephalad to the interspace between the seventh cervical and the first thoracic vertebral body NOTE: *If an MRI is not medically feasible, patients may have a CT scan with contrast

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN
* PT/PTT no greater than 1.2 times ULN

Renal:

* Not specified

Cardiac:

* No severe cardiac disease, including any of the following:

  * Uncontrolled arrhythmias or conduction defects
  * Major problems with edema (e.g., residual swelling in the legs from deep vein thrombosis)
  * Recent coronary artery disease
  * Poorly controlled hypertension (i.e., diastolic blood pressure greater than 110 mm Hg and/or systolic blood pressure greater than 180 mm Hg)

Pulmonary:

* DLCO at least 70% of predicted
* No severe pulmonary disease

Other:

* HIV negative
* No severe Cushing's syndrome
* No known allergies to any of the study drugs
* No major psychiatric illness
* No poorly controlled diabetes complicated by steroid treatment
* No other medical illness that cannot be adequately controlled or that would preclude study participation
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent antitumor chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except postmenopausal estrogen replacement therapy
* Corticosteroids at stable or decreasing dose for tumor edema allowed

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy
* No other concurrent radiotherapy (including intensity-modulated radiotherapy) to the index lesion(s)

Surgery:

* See Disease Characteristics
* No concurrent antitumor surgery

Other:

* No other concurrent investigational drugs
* No other concurrent antineoplastic drugs or therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2001-09; Primary Completion 2006-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Survival | assessed every 6 weeks for 42 weeks, then every 4 months for one year, followed by every 6 months for years 2 through 5

SECONDARY OUTCOMES:
Progression-free survival | assessed every 6 weeks for 42 weeks, then every 4 months for one year, followed by every 6 months for years 2 through 5
Time to treatment failure | assessed every 6 weeks for 42 weeks, then every 4 months for one year, followed by every 6 months for years 2 through 5
Toxicity | assessed weekly for 42 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah T. Blumenthal, MD, Study Chair — University of Utah; Alexander M. Spence, MD, Study Chair — University of Washington; Keith J. Stelzer, MD, PhD, Study Chair — Celilo Cancer Center at Mid-Columbia Medical Center
Locations (163):
- United States (163):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Banner Thunderbird Medical Center, Phoenix, Arizona
  - North Bay Cancer Center, Fairfield, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Anthony North Hospital, Westminster, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Good Samaritan Health Systems, Kearney, Nebraska
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Capital Medical Center, Olympia, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Blumenthal DT, Wade M, Rankin CJ, et al.: MGMT methylation in newly-diagnosed glioblastoma multiforme (GBM): from the S0001 phase III study of radiation therapy (RT) and O6-benzylguanine, (O6BG) plus BCNU versus RT and BCNU alone for newly diagnosed GBM. [Abstract] J Clin Oncol 24 (Suppl 18): A-1512, 2006.
- [Result] Quezado M, Ronchetti R, Rapkiewicz A, Santi M, Blumenthal DT, Rushing EJ. Chromogenic in situ hybridization accurately identifies EGFR amplification in small cell glioblastoma multiforme, a common subtype of primary GBM. Clin Neuropathol. 2005 Jul-Aug;24(4):163-9. PMID 16033132
- [Derived] Blumenthal DT, Rankin C, Stelzer KJ, Spence AM, Sloan AE, Moore DF Jr, Padula GD, Schulman SB, Wade ML, Rushing EJ. A Phase III study of radiation therapy (RT) and O(6)-benzylguanine + BCNU versus RT and BCNU alone and methylation status in newly diagnosed glioblastoma and gliosarcoma: Southwest Oncology Group (SWOG) study S0001. Int J Clin Oncol. 2015 Aug;20(4):650-8. doi: 10.1007/s10147-014-0769-0. Epub 2014 Nov 19. PMID 25407559